CLINICAL TRIAL: NCT04778215
Title: Prevention and Treatment of Low Back Pain in Young Female TeamGym Gymnasts - a Cluster Randomized Controlled Intervention Study
Brief Title: Prevention and Treatment of Low Back Pain in Young Female TeamGym Gymnasts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Marita Löfgren Harringe, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KI2009/1414-31/3; Dnr 4646/2011-631 (Other: PUL, Karolinska Institutet, Sweden)
Record Dates: First submitted 2011-08-18; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Low Back Pain
Keywords: stabilization training; abdominal hollowing; gymnastics
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): progressive, 8 week lumbar stabilizing program
  Interventions: Other: A progressive specific lumbar stabilization program
- Control group (No Intervention): Continue as usual

INTERVENTIONS:
Other: A progressive specific lumbar stabilization program — The aim of these programs is to optimize the stabilization and control of segmental motion of the lumbar spine. It is based on the draw-in action, hereafter called the abdominal hollowing, presented by Richardson and Jull (1995). The training program consists of three levels. Level 1 introduces the abdominal hollowing exercise in the prone and four-point kneeling position. Level 2 is a progression of these exercises and the gymnasts are also instructed to perform the abdominal hollowing standing on a balance board with slightly flexed knees while slowly moving the arms. Level 3 takes the training into sports specificity and the abdominal hollowing are to be held during three different basic trampette jumps with emphasis on good trunk and body control during jumping and landing.
  Other Names: Draw-in-action, abdominal hollowing, core
  Arms: Intervention group

SUMMARY:
Specific stabilization training targeting the deep trunk muscles has shown good effect in the rehabilitation of Low Back Pain (LBP) in young female TeamGym (TG) gymnasts. However, if this training can prevent LBP in this young population remains to be investigated. The aim of the present study was to investigate if a specific lumbar stabilization program can reduce and prevent LBP in young female TG gymnasts.

DETAILED DESCRIPTION:
Objectives: To study if a progressive specific lumbar stabilization program can reduce and prevent low back pain (LBP) in young female TeamGym (TG) gymnasts aged 10-16 years.

Design A cluster randomized controlled intervention study

Participants: All available competitive youth female TG teams including gymnasts aged 10-16 years, in the area of Stockholm, were invited to participate in the present study. A team consists of approximately 16 gymnasts. Fourteen out of 17 teams and a total of 258 gymnasts accepted to participate. Gymnasts and parents were informed about the study and written consent was collected. A cluster randomization process was undertaken as follows: the gymnasts in each team answered questions at inclusion and the teams were matched with respect to age, level of competition, amount of training sessions per week and reports of LBP. LBP in this study was defined as; "pain between the 12th rib and the gluteal fold". Thereafter a cluster randomization took place. This means that all gymnasts in one team were either in the control or in the intervention group. There were no differences with respect to demographic and training data and reports of LBP between the two groups at randomization. Ninety gymnasts did not report LBP at inclusion or during baseline and were included in a subgroup analysis on the preventive effect of the exercise program.

Methods Every week the gymnasts were visited by a registered physical therapist (RPT). The RPT answered questions from the gymnasts concerning injuries and collected a weekly-based questionnaire. The gymnasts in the intervention group were instructed to perform an eight-week progressive specific lumbar stabilization program, implemented in the warm-up at every training session. The gymnasts answered a weekly based questionnaire regarding training and LBP during the intervention period, and thereafter a questionnaire at 3-, 6- and 12 months follow-up. The gymnasts and the coaches were also instructed to continue with the lumbar stabilization program after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* female TeamGym teams, aged 10-16 years, in the Stockholm area
* competing at national or international level

Exclusion Criteria:

* male TeamGym gymnasts
* female TeamGym teams on a regional competitive level

Ages: 10 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 258 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Weekly prevalence of LBP from baseline to end of the intervention program | 3 months
  Number of gymnasts reporting LBP/ Total number of gymnasts' reports; comparing the intervention and control group
Weekly prevalence of SLBP (Substantial LBP) from baseline to end of the intervention program | 3 months
  Number of gymnasts reporting LBP 3 days or more or modification of participation (SLBP)/ Total number of gymnasts' reports; comparing the intervention and control group
Prevalence of LBP at 3-, 6- and 12 months follow up | 18 months
  Number of gymnasts reporting LBP/ Total number of gymnasts' reports; comparing the intervention and control group

SECONDARY OUTCOMES:
Change of Intensity and prevalence of LBP in gymnasts that report SLBP at the start of the study - from baseline to end of intervention, and at 3-, 6- and 12 months follow-up | 18 months
  Subgroup analysis including gymnasts with SLBP at the start of the study; comparing intervention and control group
Prevention of LBP evaluated after intervention and at 3-, 6- and 12 months | 18 months
  Subgroup analysis including gymnasts with no previous LBP at the start of the study; comparing intervention and control group

CONTACTS AND LOCATIONS:
Overall Officials: Marita L Harringe, PhD,RPT, Study Director — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Department of Molecular Medicine and Surgery, Stockholm Sports Trauma Research Center, Stockholm, Sweden